CLINICAL TRIAL: NCT03132714
Title: Local Effect of Periodontal Debridement Associated With Different Systemic Antibiotic Protocols and Single or Repeated Application of Photodynamic Therapy to Treat Generalized Aggressive Periodontitis: Randomized Controlled Clinical Trial
Brief Title: Periodontal Debridement Associated With Systemic Antibiotics and Single/Repeated PDT to Treat Aggressive Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, PhD Adjunct professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rPDT&antibioticsCFA
Record Dates: First submitted 2017-04-23; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Aggressive Periodontitis, Generalized
Keywords: Full-mouth ultrasonic debridement; Clarithromycin; Amoxicillin; Metronidazole; Antimicrobial therapy; Photodynamic therapy; Low-level laser therapy
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Periodontal Debridement; Amoxicillin; Metronidazole; Clarithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- PD + (AMX + MET) (Active Comparator): periodontal pockets that will receive full-mouth ultrasonic debridement associated with systemic Amoxicillin 500 mg + Metronidazole 400 mg
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Amoxicillin 500mg; Drug: Metronidazole 400mg
- PD + CLM (Active Comparator): periodontal pockets that will receive full-mouth ultrasonic debridement associated with systemic clarithromycin 500 mg
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Clarithromycin 500mg
- PD + (AMX + MET) + sPDT (Active Comparator): periodontal pockets that will receive full-mouth ultrasonic debridement associated with systemic Amoxicillin 500 mg + Metronidazole 400 mg and single application of PDT
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Amoxicillin 500mg; Drug: Metronidazole 400mg; Procedure: Single application of PDT
- PD + CLM + sPDT (Active Comparator): periodontal pockets that will receive full-mouth ultrasonic debridement associated with systemic Clarithromycin 500 mg and single application of PDT
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Clarithromycin 500mg; Procedure: Single application of PDT
- PD + (AMX + MET) + rPDT (Active Comparator): periodontal pockets that will receive full-mouth ultrasonic debridement associated with systemic Amoxicillin 500 mg + Metronidazole 400 mg and repeated application of PDT
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Amoxicillin 500mg; Drug: Metronidazole 400mg; Procedure: Repeated application of PDT
- PD + CLM + rPDT (Active Comparator): periodontal pockets that will receive full-mouth ultrasonic debridement associated with systemic Clarithromycin 500 mg and repeated application of PDT
  Interventions: Procedure: Full-mouth ultrasonic debridement; Drug: Clarithromycin 500mg; Procedure: Repeated application of PDT

INTERVENTIONS:
Procedure: Full-mouth ultrasonic debridement — Full-mouth ultrasonic debridement will be performed in order to treat diseased sites
  Other Names: Periodontal debridement
Drug: Amoxicillin 500mg — Administration of Amoxicillin 500mg tid for 7 days
  Other Names: Amoxil
  Arms: PD + (AMX + MET); PD + (AMX + MET) + rPDT; PD + (AMX + MET) + sPDT
Drug: Metronidazole 400mg — Administration of Metronidazole 400mg tid for 7 days.
  Other Names: Flagyl
  Arms: PD + (AMX + MET); PD + (AMX + MET) + rPDT; PD + (AMX + MET) + sPDT
Drug: Clarithromycin 500mg — Administration of Clarithromycin 500mg bid for 7 days
  Other Names: Biaxin
  Arms: PD + CLM; PD + CLM + rPDT; PD + CLM + sPDT
Procedure: Single application of PDT — Single application of photodynamic therapy (PDT) at day 0.
  Arms: PD + (AMX + MET) + sPDT; PD + CLM + sPDT
Procedure: Repeated application of PDT — Repeated application of photodynamic therapy (PDT) at 0, 1, 2, 7 and 14 days post-operatively.
  Arms: PD + (AMX + MET) + rPDT; PD + CLM + rPDT

SUMMARY:
The aim of this project is to compare the efficacy and the local effect of the association of single or repeated application of photodynamic therapy (PDT) with antibiotic agents using Amoxicillin + Metronidazole or Clarithromycin in the treatment of patients with Generalized Aggressive Periodontitis (GAgP).

DETAILED DESCRIPTION:
The study methodology is according to CONSORT-STATEMENT 2010 and SPIRIT 2013 for randomized controlled clinical trials.

Study Design

The study is designed as a prospective, interventional, parallel, blinded, randomized, controlled clinical trial aimed to compare the efficacy and the local effect of the association of single or repeated application of photodynamic therapy (PDT) with antibiotic agents using Amoxicillin + Metronidazole or Clarithromycin in the treatment of patients with Generalized Aggressive Periodontitis (GAgP).

Source of data

The population of this study will be recruited among patients referred to the Science and Technology Institute (ICT) - São José dos Campos, College of Dentistry. Each one of 46 patients will have three pockets with probing depth and loss of clinical attachment level ≥5 mm and bleeding on probing not located at furcation sites randomly chosen.

Power calculation

A population of 46 patients (138 periodontal pockets, 3 per patient) that meet the pre-established criteria will be considered. Considering α = 5% and a β = 5% to detect a difference of 1 mm between groups in probing depth reduction of pockets ≥5 mm, for a standard deviation of 0.8 mm, 14 patients will be needed in each group. With a sample of 46 patients (138 pockets), the study will have a power greater than 95%.

Clinical Parameters

All clinical parameters will be assessed by a single blinded, trained and calibrated examiner (CFA) before periodontal therapy (baseline) and at 3 and 6 months after using a manual probe. Measurements will be done at six sites per tooth (mesiobuccal, buccal, disto-buccal, distolingual, lingual, and mesiolingual) in all teeth, except third molars.

The following clinical parameters will be evaluated: 1) Full-mouth plaque index (FMPI); 2) Bleeding on probing (BoP); 3) Probing depth (PD): distance from the bottom of sulcus/pocket to gingival margin; 4) Gingival recession (GM): distance from the free gingival margin to cement-enamel junction (CEJ); 5) Clinical attachment level (CAL): distance from bottom of sulcus/pocket to the CEJ. The CEJ will be identified by careful probe on cervical area.

Calibration and Randomization

Initially, a total of ten patients presenting with GAgP will be selected. The designated examiner (CFA) will measure CAL and PD in all patients twice within 24 hours, with an interval of ≥ 1 hour between examinations. Then, the measures will be submitted to intraclass correlation test and the examiner will be judged calibrated if reaches 90% agreement.

Patients will be allocated into two antibiotic groups (that will receive Amoxicillin + Metronidazole or Clarithromycin) according to a computer-generated list. The allocation will be implemented by an investigator (NCCS) who was not directly involved in the examination or treatment procedures. All medication will be prepared and encased in identical opaque coded bottles by a compounding pharmacy. The same person outside the project will generate a random sequence regarding the type of PDT application for each patient, for the three previously selected pockets (single or repeated application of PDT or control), which will be revealed shortly after the periodontal debridement session.

Treatment Protocols

All patients will be treated with periodontal therapy through of the one-stage, full mouth, ultrasonic debridement (FMUD). In a single session, patients will receive local anesthesia and periodontal debridement with ultrasound equipment (Cavitron - Dentsply EUA) and subgingival tips (UI25KSF10S, Hu-Friedy). All diseased sites will be instrumented in this one session. The debridement session will be performed by a single experienced and trained periodontist (NA), different from the examiner (ca). Immediately before the mechanical therapy, patients will be allocated in one of the two treatment protocols: Clarithromycin (CLM) group (n = 22): FMUD + CLM 500 mg bid, for 7 days or Amoxicillin (AMX) + metronidazole (MET) group (n = 22): FMUD + (AMX 500 mg tid + MET 400 mg tid, both for 7 days. All patients will start taking the pills immediately before the FMUD session.

After periodontal debridement (PD), two periodontal pockets from each patient will receive the proposed PDT protocols to assist the decontamination of diseased sites. One pocket will receive a single application of PDT (sPDT) (baseline only) and the other will receive repeated application of PDT (rPDT). After subgingival irrigation with saline solution to wash the pocket, the photosensitizer (methylene blue 10 mg / mL) will be applied to the bottom of the pocket by buccal side until it is completely filled. After one minute, the pocket will be washed with water and exposed to low-level laser (TheraLase - Brazil), with a corresponding optical fiber of 600 um diameter, which will be inserted into the pocket. A 660 nm wavelength with a power of 60 milliwatts and a dose of 129 J / cm2 will be used for one minute. The same procedure will be repeated by lingual site, totaling two minutes of application per pocket. The repeated application protocol will consist of 5 applications on different days, performed on the day of periodontal treatment (baseline - 0), 1, 2, 7 and 14 days after. Thus, the following comparative groups will be formed, totaling 138 pockets:

PD + (AMX + MET) (n = 23): periodontal pockets that will receive periodontal debridement associated with Amoxicillin + Metronidazole;

PD + CLM (n = 23): periodontal pockets that will receive periodontal debridement associated with the use of Clarithromycin;

PD + (AMX + MET) + sPDT (n = 23): periodontal pockets that will receive periodontal debridement associated with Amoxicillin + Metronidazole and single application of PDT; PD + CLM + sPDT (n = 23): periodontal pockets that will receive periodontal debridement associated with the use of Clarithromycin and single application of PDT;

PD + (AMX + MET) + rPDT (n = 23) : periodontal pockets that will receive periodontal debridement associated with Amoxicillin + Metronidazole and repeated application of PDT;

PD + CLM + rPDT (n = 23): periodontal pockets that will receive periodontal debridement associated with Clarithromycin and repeated application of PDT

Statistical analysis

Mean and standard deviation will be calculated for each parameter. The normal distribution of the data will be analyzed by Shapiro-Wilk test. Data from clinical measurements will be subjected to analysis of variance (repeated measures) for inter and intra-group comparison.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GAgP (Armitage, 1999; American Academy of Periodontology, 2015);
* presence of ≥20 teeth, excluding third molars and teeth indicated for extraction;
* presence of ≥6 sites presenting PD ≥5 mm with bleeding on probing and ≥2 sites with PD ≥7 mm (including incisors and first molars, in addition to two other non-contiguous teeth between them);
* presence of three non-adjacent periodontal pockets with probing depth ≥5 mm and bleeding on probing not located in furcation area;
* good general health (ASA I/II);
* 18-35 years old;
* agree to participate in the study and sign a written consent (Resolution # 196 of October 1996 and the Brazilian Professional Code of Dental Ethics - 179/93).

Exclusion Criteria:

* pregnant or nursing;
* suffer from any systemic disease (e.g. cardiovascular, diabetes, blood dyscrasias, immunodeficiency, etc - ASA III/IV/V);
* antimicrobials or anti-inflammatory drugs in the previous 6 months;
* periodontal treatment within the last 12 months;
* smoke ≥10 cigarettes/day;
* reported allergy to amoxicillin, metronidazole or clarithromycin;
* required antibiotic prophylaxis;
* current use of any medication that could interfere with periodontal response were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in Probing Depth (PD) | 0, 3 and 6 post-operatively
  Evaluate the difference between baseline and 6 months PD measures.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, DDS, PhD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- College of Dentistry - São José dos Campos, São Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lulic M, Leiggener Gorog I, Salvi GE, Ramseier CA, Mattheos N, Lang NP. One-year outcomes of repeated adjunctive photodynamic therapy during periodontal maintenance: a proof-of-principle randomized-controlled clinical trial. J Clin Periodontol. 2009 Aug;36(8):661-6. doi: 10.1111/j.1600-051X.2009.01432.x. Epub 2009 Jun 25. PMID 19563331